CLINICAL TRIAL: NCT04210427
Title: Cystic Fibrosis and Gut Dysmotility: The Effect of Polyethylene Glycol (PEG) on Intestinal Transit
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Dhiren Patel, MD, Associate Professor, St. Louis University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 30114
Record Dates: First submitted 2019-12-18; First posted 2019-12-24 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-07

CONDITIONS: Cystic Fibrosis Gastrointestinal Disease
Keywords: Cystic Fibrosis; Gut Dysmotility; Polyethylene Glycol
MeSH Terms: conditions — Cystic Fibrosis | interventions — polyethylene glycol 3350

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Intervention with polyethylene glycol & SmartPill (Experimental): Patients will ingest a Smart pill to obtain baseline motility within the GI lumen. All patients will undergo intervention with taking polyethylene glycol (PEG) or Miralax (brand name) 17 grams once daily. After two weeks of therapy, the patient will repeat the motility survey and again ingest a smart pill to assess the change in motility symptoms while on therapy.
  Interventions: Drug: Polyethylene Glycol 3350; Device: SmartPill Motility System & PillCam Patency Capsule

INTERVENTIONS:
Drug: Polyethylene Glycol 3350 — All patients will undergo intervention with taking polyethylene glycol (PEG) or Miralax (brand name) 17 grams once daily for total of 2 weeks.
Device: SmartPill Motility System & PillCam Patency Capsule — Patients will ingest a Smart pill to obtain baseline motility within the GI lumen. After two weeks of therapy, the patient will repeat the motility survey and again ingest a smart pill to assess the change in motility symptoms while on therapy.

SUMMARY:
The investigators will recruit 15 patients with cystic fibrosis 18 years of age and older who present with constipation. The investigators will assess baseline motility symptoms with a survey. Patients will then ingest a SmartPill (trademark) to obtain baseline motility within the GI lumen. All patients will undergo intervention with taking polyethylene glycol (PEG) or Miralax (brand name) 17 grams once daily. After two weeks of therapy, the patient will repeat the motility survey and again ingest a smart pill to assess the change in motility symptoms while on therapy.

DETAILED DESCRIPTION:
Background:

Cystic Fibrosis (CF) is an autosomal recessive disorder involving mutation of the cystic transmembrane conductance regulator (CFTR) protein. The consequences of this genetic mutation leads to dysregulated epithelial fluid transportation. Abnormalities of the CFTR protein have multisystem motility complications - it affects primarily the lungs, pancreas, vas deferens, and the gastrointestinal (GI) tract. Cystic Fibrosis causes multiple issues in the GI tract. The CFTR protein is expressed throughout the GI tract at the apical enterocyte membrane. Per recent studies, it has the highest concentration in the duodenum and decreases as the small bowel terminates into the large intestine. Patients often experience symptoms secondary to dysmotility from abnormal salt and water regulation into the gastrointestinal lumen. Cystic Fibrosis patients are at risk for small intestinal bacterial overgrowth (SIBO), intestinal dysbiosis, inflammation, distal intestinal obstruction syndrome (DIOS), constipation, and postprandial delayed gastric emptying.

Multiple studies have been done to evaluate gastrointestinal motility in the CF patients. One study reviewed gastric muscle rhythms in CF patients via pre and post-prandial electrogastrography (EGG) and found postprandial bradygastria. Patients had symptom improvement with initiation of cisapride however this drug is not FDA approved in different continents. Another study researched GI transit times via the magnet-based motility tracking system and found increased transit in the upper small intestine compared to control populations. Overall, CF patients were found to have delayed small intestine transit time with the magnetic pill reaching the cecum in only 2 of 10 CF patients in a 7 hour period compared to 14 of 16 control patients. Hydrogen Breath tests have diagnosed SIBO in CF patients however overall delay in intestinal transit affect interpretation of results. Empiric treatment with antibiotics or laxatives is recommended with some improvement in patient symptoms. Mouse studies have shown that use of Miralax (brand name) or polyethylene glycol (PEG) laxative decreased bacterial overgrowth in 90% of Cystic Fibrosis mice. Further studies showed that daily PEG use decreases positive breath tests in a small study of CF patients. While there have been multiple studies showing symptomatic improvement of SIBO and DIOS with PEG and/or other laxative agents, none have measured whether or not these medications improve intestinal transit time. The aim of this research project is to evaluate total intraluminal transit time in CF patients and the effects of PEG on transit time and patient symptoms.

Study Description:

This is a prospective cohort study. This is an investigator initiated study. Once enrolled, patients will spend a total of 4 weeks in the study. All participants will receive the intervention. There will be no randomization in this study.

Information pulled from the patient's medical record includes the patient's name, medical record number, date of birth, cystic fibrosis genotype, medication list, and medical history.

Study Procedures:

1. Initial recruiting visit: Informed consent to participate in the research study will be obtained.The patient will need to have a 2 week washout period where all non-essential medications that alter gut motility are temporarily stopped. The medications withheld will be at the discretion of the physician.This list will be provided to the patient. The patients on pancreatic enzyme replacement must remain on this as to not affect study outcomes.
2. Second visit: The patient will complete Rome IV Diagnostic Questionnaire (R4DQ) for Functional Gastrointestinal Disorders in Adults (FGIDs). This Questionnaire is considered a research procedure. Once procedural informed consent is obtained, the patient will be fitted for the recorder and ingest the SmartPill. The patient will return the receiver up to seven days after the capsule was ingested.The SmartPill is considered a research procedure. If the SmartPill is not excreted after day 7, the patient will obtain an outpatient abdominal X-ray to determine if the SmartPill device is retained in the intestines. A pregnancy test will be performed prior to any potential radiation exposure for female patients of child-bearing ages, 13-50 years old. The X-ray, if completed, is considered a research procedure.

   **If there is concern the SmartPill may be retained in the intestine, the patient may be asked to take a Patency agile capsule. This will require the patient to obtain a abdominal X-ray 24 hours after ingestion as an outpatient to localize the capsule's location. This is considered standard of care.
3. Study period (two weeks): After 7 days, the patient will begin intervention with polyethylene glycol (PEG) 17 g therapy for total of 2 weeks. If persistent symptoms (no bowel movements in > 24 hours, abdominal pain, straining, bloating), then the patient can increase to 17 g twice daily. The patient will call the office after 1 week to determine if step up to twice daily therapy is warranted.

   The patients will receive a log to record time of PEG ingestion, if PEG was taken with meals, a log of other medications taken during the intervention timeline, and recording symptoms of constipation. Patients will be advised to avoid non-essential drugs that can alter gut motility (see attached list found on the patient log) during the treatment period. The study drug is considered standard of care procedure.
4. Third visit: Two weeks following initiation of therapy, the patient will repeat the Rome IV Diagnostic Questionnaire for Adult FGIDs (R4DQ) and ingest the second SmartPill to assess for change in gut motility. Procedural informed consent will be obtained prior the questionnaire and ingestion of the SmartPill. This Questionnaire and SmartPill device is considered a research procedure. The patient will return the receiver up to seven days after the capsule was ingested.The SmartPill is considered a research procedure. If the SmartPill is not excreted after day 7, the patient will obtain an outpatient abdominal XRay to determine if the SmartPill device is retained in the intestines. A pregnancy test will be performed prior to any potential radiation exposure for female patients of child-bearing ages, 13-50 years old.The X Ray, if completed, is considered a research procedure.

   **If there is concern the SmartPill may be retained in the intestine, the patient may be asked to take a Patency agile capsule. This will require the patient to obtain a abdominal X Ray 24 hours after ingestion as an outpatient to localize the capsule's location. This is considered standard of care.
5. Fourth visit: The patient will return the recorder equipment for analysis and will complete a post study questionnaire and undergo review of their therapy log detailing how the medication was taken. This Questionnaire is considered a research procedure.

The subject participation in the study ends at this point.

ELIGIBILITY:
Inclusion Criteria:

* previously diagnosed with CF confirmed with genetic mutations consistent with CF
* greater than 18 years old who chose to participate in the research study
* have symptoms of constipation (constipation will be defined as stool frequency less than three times per week, Bristol stool scale form 1-2 in >25% of stools, and/or the sensation of incomplete evacuation, manual maneuvers to facilitate stools, and the sensation of blockage)

The patients enrolled are allowed to be on CFTR modulating drugs and/or receiving enteral feeding.

Exclusion Criteria:

* minors (<18 years old)
* active nicotine use or patients on nicotine replacement
* history of abdominal surgery (surgeries involving gastrointestinal luminal resection) ie small bowel or colonic resection that increases risk of post-operative strictures or narrowing of the lumen. Surgeries such as Nissen fundoplication, gastrostomy tube placement, gynecologic surgeries, appendectomy, and/or cholecystectomy are not excluded from this study.
* history of lung transplantation or pancreas transplant
* BMI >40
* pregnancy (this will be screened via urine pregnancy test)
* incarcerated persons
* patients with DIOS (distal intestinal obstructive syndrome)
* patients with known hypersensitivity to PEG
* persons unable to remain off the contraindicated medications.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dhiren Patel, MD, Principal Investigator — St. Louis University
Locations (2):
- United States (2):
  - SSM Health Cardinal Glennon Children's Hosptial, St Louis, Missouri
  - SSM Health Saint Louis University Hosptial, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Corral JE, Dye CW, Mascarenhas MR, Barkin JS, Salathe M, Moshiree B. Is Gastroparesis Found More Frequently in Patients with Cystic Fibrosis? A Systematic Review. Scientifica (Cairo). 2016;2016:2918139. doi: 10.1155/2016/2918139. Epub 2016 May 30. PMID 27313953
- [Result] Hedsund C, Gregersen T, Joensson IM, Olesen HV, Krogh K. Gastrointestinal transit times and motility in patients with cystic fibrosis. Scand J Gastroenterol. 2012 Sep;47(8-9):920-6. doi: 10.3109/00365521.2012.699548. Epub 2012 Jul 2. PMID 22746323
- [Result] Bentur L, Hino B, Shamir R, Elias N, Hartman C, Eshach-Adiv O, Berkowitz D. Impaired gastric myolectrical activity in patients with cystic fibrosis. J Cyst Fibros. 2006 Aug;5(3):187-91. doi: 10.1016/j.jcf.2006.03.003. Epub 2006 Apr 19. PMID 16627012
- [Result] Dorsey J, Gonska T. Bacterial overgrowth, dysbiosis, inflammation, and dysmotility in the Cystic Fibrosis intestine. J Cyst Fibros. 2017 Nov;16 Suppl 2:S14-S23. doi: 10.1016/j.jcf.2017.07.014. PMID 28986022
- [Result] Schappi MG, Roulet M, Rochat T, Belli DC. Electrogastrography reveals post-prandial gastric dysmotility in children with cystic fibrosis. J Pediatr Gastroenterol Nutr. 2004 Sep;39(3):253-6. doi: 10.1097/00005176-200409000-00005. PMID 15319624
- [Result] Xu RB, Bhuyan RR, Edwards JR. Staged Bentall procedure and extra-anatomical repair of coarctation of aorta. ANZ J Surg. 2016 Apr;86(4):310-1. doi: 10.1111/ans.12666. Epub 2014 May 29. No abstract available. PMID 24891257
- [Result] Palsson OS, Whitehead WE, van Tilburg MA, Chang L, Chey W, Crowell MD, Keefer L, Lembo AJ, Parkman HP, Rao SS, Sperber A, Spiegel B, Tack J, Vanner S, Walker LS, Whorwell P, Yang Y. Rome IV Diagnostic Questionnaires and Tables for Investigators and Clinicians. Gastroenterology. 2016 Feb 13:S0016-5085(16)00180-3. doi: 10.1053/j.gastro.2016.02.014. Online ahead of print. PMID 27144634

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention With Polyethylene Glycol & SmartPill
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients with GI symptoms and Cystic Fibrosis.
Groups:
- Intervention With Polyethylene Glycol & SmartPill: Patients will ingest a Smart pill to obtain baseline motility within the GI lumen. All patients will undergo intervention with taking polyethylene glycol (PEG) or Miralax (brand name) 17 grams once daily. After two weeks of therapy, the patient will repeat the motility survey and again ingest a smart pill to assess the change in motility symptoms while on therapy.
  Polyethylene Glycol 3350: All patients will undergo intervention with taking polyethylene glycol (PEG) or Miralax (brand name) 17 grams once daily for total of 2 weeks.
  SmartPill Motility System & PillCam Patency Capsule: Patients will ingest a Smart pill to obtain baseline motility within the GI lumen. After two weeks of therapy, the patient will repeat the motility survey and again ingest a smart pill to assess the change in motility symptoms while on therapy.
  Total of 3 patients participated.
Arm/Group | Intervention With Polyethylene Glycol & SmartPill
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Change is Being Assessed: Total Intestinal Transit Time at Baseline and Two Weeks Following Initiation of Therapy
Description: Total intestinal transit time will be measured from the time of ingestion to time of expulsion of smartpill. Unit of measurement will be hours.
Time Frame: Change is being assessed: total intestinal transit time (measured in hours) at baseline and two weeks following initiation of therapy with PEG
Population: Adult patients with Cystic Fibrosis with gastrointestinal symptoms.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Intervention With Polyethylene Glycol & SmartPill
Number analyzed (Participants) | 3
hours
  total intestinal transit time - baseline | 41 (13)
  total intestinal transit time-2 weeks after PEG therapy | 42 (14)

2. Primary Outcome: Number of Participants With IBS at Baseline and 2 Weeks Post Baseline
Description: Subjective assessment for abdominal symptoms with ROME questionnaire. Note that the outcome of these questionnaire is IBS present or absent.Rome 4 is a self-report integrated questionnaire in adults (R4DQ), including alarm symptoms or red flags.
  ROME 4 IBS present if:
  Recurrent abdominal pain on average at least 1 day/week in the last 3 months, associated with two or more of the following criteria:
  Related to defecation Associated with a change in frequency of stool Associated with a change in form (appearance) of stool
  Criteria fulfilled for the last 3 months with symptom onset at least 6 months prior to diagnosis.
  Rome 4 IBS absent if not fulfilled as above.
Time Frame: Baseline and 2 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Intervention With Polyethylene Glycol & SmartPill: Patients will ingest a Smart pill to obtain baseline motility within the GI lumen. All patients will fill out ROME questionnaire before PEG or Smartpill. All patients will undergo intervention with taking polyethylene glycol (PEG) or Miralax (brand name) 17 grams once daily. After two weeks of therapy, the patient will repeat the ROME survey to evaluate IBS and again ingest a smart pill to assess the change in motility while on therapy.
  Polyethylene Glycol 3350: All patients will undergo intervention with taking polyethylene glycol (PEG) or Miralax (brand name) 17 grams once daily for total of 2 weeks.
  SmartPill Motility System & PillCam Patency Capsule: Patients will ingest a Smart pill to obtain baseline motility within the GI lumen. After two weeks of therapy, the patient will repeat the motility survey and again ingest a smart pill to assess the change in motility symptoms while on therapy.
  Total of 3 patients participated.
Arm/Group | Intervention With Polyethylene Glycol & SmartPill
Number analyzed (Participants) | 3
Participants
  ROME 4- IBS present at baseline | 3
  ROME 4- IBS absent at baseline | 0
  ROME 4 IBS present at 2 weeks after PEG/Smartpill | 3
  ROME 4 IBS absent at 2 weeks after PEG/Smartpill | 0

ADVERSE EVENTS:
Time Frame: Overall time frame for the study: 2 years 4 months. Adverse events were recorded during and after the use of smartpill up to 2 weeks. For all three participants the period of collection of adverse event was 8 weeks. Informed consent and Baseline Rome questionnaire for GI symptoms - Week 1, Administer smart pill - Week 3,Collect transit time and related data - Week 4,Start Polyethylene Glycol - Week 5,Administer SmartPill again in 2 weeks - Week 7, Repeat the questionnaire - week 8
Groups:
- Intervention With Polyethylene Glycol & SmartPill: Patients will ingest a Smart pill to obtain baseline motility within the GI lumen. All patients will undergo intervention with taking polyethylene glycol (PEG) or Miralax (brand name) 17 grams once daily. After two weeks of therapy, the patient will repeat the motility survey and again ingest a smart pill to assess the change in motility symptoms while on therapy.
  Polyethylene Glycol 3350: All patients will undergo intervention with taking polyethylene glycol (PEG) or Miralax (brand name) 17 grams once daily for total of 2 weeks.
  SmartPill Motility System & PillCam Patency Capsule: Patients will ingest a Smart pill to obtain baseline motility within the GI lumen. After two weeks of therapy, the patient will repeat the motility survey and again ingest a smart pill to assess the change in motility symptoms while on therapy.
  We did not collect the outcome details due to not adequate patients' participation. No adverse events were reported throughout the study.
Arm/Group | Intervention With Polyethylene Glycol & SmartPill
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan: Main protocol and analysis plan (2023-06-08): https://cdn.clinicaltrials.gov/large-docs/27/NCT04210427/Prot_SAP_001.pdf